CLINICAL TRIAL: NCT01180413
Title: Effects of Intensive Vasodilating add-on Therapy on Peripheral Vascular Resistance and Coronary Flow Reserve in Patients With Essential Hypertension
Brief Title: Intensive Vasodilator Therapy in Patients With Essential Hypertension
Acronym: Vasomore
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Morten Engholm Pedersen, MD/PhD-Student, Aarhus University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26169
Record Dates: First submitted 2010-08-11; First posted 2010-08-12 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Essential Hypertension; High Blood Pressure
Keywords: Inward eutrophic remodelling
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — Amlodipine; Ramipril; lercanidipine; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vasodilatory (Experimental): Patients in this arm will receive intensive vasodilatory treatment
  Interventions: Drug: Amlodipine; Drug: Ramipril; Drug: Lercanidipine; Drug: Losartan

INTERVENTIONS:
Drug: Amlodipine — 5 mg per day for 6 months as add-on to original ongoing antihypertensive treatment
  Other Names: Amlodipin
Drug: Ramipril — 5 mg per day for the first to weeks as add-on to original ongoing antihypertensive treatment. Then upward adjustment to 10 mg per day for 6 months if no intolerable side effects are experienced.
Drug: Lercanidipine — Up to 20 mg per day for 6 months as add-on to original ongoing antihypertensive treatment
Drug: Losartan — Up to 100 mg per day for 6 months as add-on to original ongoing antihypertensive treatment

SUMMARY:
The purpose of this study is to determine whether add-on of intensive vasodilator therapy can improve the coronary perfusion and reduce the total peripheral resistance in patients with ongoing treatment for essential hypertension.

DETAILED DESCRIPTION:
Morphological changes are observed in the microvasculature of patients with essential hypertension. The lumen diameter is reduced in resistance arteries, but with no change in vessel cross-sectional area or wall mass. These structural changes are termed inward eutrophic remodelling and results in an increased wall:lumen ratio, caused by rearrangement of cell matrix and not by hypertrophy of smooth muscle cells in the vascular wall as observed in secondary forms of hypertension. The morphological changes also occur in the coronary arteries and cause a reduction in the ability to increase coronary perfusion as response to increased cardiac work. This is observed as a reduced coronary flow reserve in patients with sustained hypertension.

Two recently published clinical studies associates an increase in media:lumen ratio with an increased risk of cardiovascular events, and it therefore seems beneficial to normalize the vascular structure in patients with essential hypertension. It has previously been demonstrated that reversion of vascular remodelling and thereby normalization of the vascular structure, requires vasodilatation and not just blood pressure reduction, suggesting that patients with essential hypertension can benefit from antihypertensive treatment aimed to induce vasodilatation.

The purpose of this study is to determine whether add-on of intensive vasodilator therapy can improve the coronary perfusion (coronary flow reserve) and reduce the total peripheral resistance in patients with ongoing treatment for essential hypertension. We also aim to investigate whether changes in coronary flow reserve correlates better to changes in total peripheral resistance than changes in blood pressure. Particularly we aim to study if patients with high total peripheral resistance, despite blood pressure control, can benefit from intensive vasodilating therapy.

ELIGIBILITY:
Inclusion Criteria:

* Ongoing antihypertensive treatment for >3 months
* Blood pressure >120/75 during antihypertensive treatment
* Ejection fraction > 45%

Exclusion Criteria:

* Blood pressure >160/100
* Pregnancy
* fertile women not using safe contraceptives
* known secondary hypertension
* valvular disease of haemodynamic significance
* known endocrine disease, nephropathy or hepatic disease
* present malignant disease
* known psychiatric disease
* abnormal lab tests of clinical significance
* known allergy to any study medication
* body mass index > 35
* Ongoing antihypertensive treatment with a combination of ACE-inhibitor and Calcium antagonist.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Coronary Flow Reserve | 6 months
  Determined by echocardiography

SECONDARY OUTCOMES:
Puls Wave Velocity | 6 months
Left ventricular mass | 6 months
  Determined with echocardiography
Blood Pressure | 6 months
  Ambulatory Blood Pressure
Peripheral Vascular Resistance | 6 months
  By Innocor
Minimal forearm vascular resistance | 6 months
  By pletysmography

CONTACTS AND LOCATIONS:
Overall Officials: Morten Engholm Pedersen, MD, Principal Investigator — Aarhus University and Aarhus University Hospital; Ole Norling Mathiasen, MD, PhD, Study Director — Aarhus University and Aarhus University Hospital; Niels Henrik Buus, DMSc, Study Director — Aarhus University and Aarhus University Hospital; Ashkan Eftekhari, MD, PhD, Principal Investigator — Aarhus University and Aarhus University Hospital
Locations (1):
- Aarhus University Hospital - dept. cardiology (A), Aarhus, Denmark